CLINICAL TRIAL: NCT05228223
Title: Comparison of Sugammadex and Sugammadex-neostigmine Combination in the Antagonism of Moderate Neuromuscular Block Induced by Rocuronium: A Prospective Randomized Cotrolled Study
Brief Title: Comparison of Sugammadex and Sugammadex-neostigmine Combination in the Antagonism of Moderate Neuromuscular Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: E1-21-1914
Record Dates: First submitted 2021-09-19; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Residual Neuromuscular Block; Neuromuscular Blockade Monitoring
Keywords: Sugammadex; Neostigmine; Neuromuscular Blockade Monitoring; Postoperative Nausea and Vomiting; Delayed Emergence from Anesthesia; Postoperative Complications; Rocuronium; Residual Neuromuscular Block
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Postoperative Nausea and Vomiting; Postoperative Complications | interventions — Neuromuscular Monitoring; Sugammadex

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled double blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group S (Active Comparator): Patients reversed with Sugammadex 2mg/kg after TOF count is 1-2.
  Interventions: Diagnostic Test: Neuromuscular monitoring; Other: reverse of NMB with sugammadex
- Group SN1 (Active Comparator): Patients reversed with Sugammadex 1mg/kg + Neostigmin 0.02 mg/kg after TOF count is 1-2.
  Interventions: Diagnostic Test: Neuromuscular monitoring; Other: reverse of NMB with Sugammadex and neostigmin low dose
- Grup SN2 (Active Comparator): Patients reversed with sugammadex 1.5 mg/kg + Neostigmin 0.02 mg/kg after TOF count is 1-2.
  Interventions: Diagnostic Test: Neuromuscular monitoring; Other: reverse of NMB with Sugammadex and neostigmin high dose

INTERVENTIONS:
Diagnostic Test: Neuromuscular monitoring — TOF monitoring
Other: reverse of NMB with sugammadex — Patients reversed with Sugammadex 2mg/kg after TOF count is 1-2.
  Arms: Group S
Other: reverse of NMB with Sugammadex and neostigmin low dose — Patients reversed with Sugammadex 1mg/kg + Neostigmin 0.02 mg/kg
  Arms: Group SN1
Other: reverse of NMB with Sugammadex and neostigmin high dose — patients reversed with sugammadex 1.5 mg/kg + Neostigmin 0.02 mg/kg
  Arms: Grup SN2

SUMMARY:
In this prospective randomized controlled study the investigators compare the sugammadex-neostigmine combination and single dose sugammadex in terms of side effects and cost for the antagonism of moderate neuromuscular block induced by rocuronium.

DETAILED DESCRIPTION:
Sugammadex is a novel drug used to reverse neuromuscular blockade. It shows its effect by binding with steroid neuromuscular agents at a ratio of 1:1. Compared to anticholinesterase and other neuromuscular reverse agents, sugammadex shows less cholinergic side effects and less residual muscle relaxation. Besides all these, sugammadex reverses neuromuscular blockade very quickly. In addition to these benefits, it has side effects such as hypersensitivity and this side effect can be seen more at high doses. In addition, sugammadex is more costly than other neuromuscular reverse agents.

In this prospective randomized controlled study the investigators compare the sugammadex-neostigmine combination and single dose sugammadex in terms of side effects and cost for the antagonism of moderate neuromuscular block induced by rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* elective general anesthesia
* Female gender
* Between the ages of 18-65

Exclusion Criteria:

* ASA ≥ 3
* Pregnancy
* Contraindication to use of anesthetic drugs
* Kidney failure
* Liver failure
* Heart failure
* BMI <18 and BMI > 35 kg/m2
* anticipated difficult airway
* neuromuscular disease
* Use of drugs that impair neuromuscular transmission
* Patients who develop unexpected massive hemorrhage
* Those who do not have the ability to read, understand and sign the consent form
* Refusal of patient

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Residual curarization rate | through study completion an average of 3 months
  Pecents of Patients TOFR<0.9
SPO2 | through study completion an average of 3 months
  peripheric oxygen saturation
MAP | through study completion an average of 3 months
  Mean arterial pressure
HR | through study completion an average of 3 months
  Heart Rate

SECONDARY OUTCOMES:
PONV | through study completion an average of 3 months
  Postoperative nausea and vomiting
Time to Return of bowel movements | through study completion an average of 3 months
  when patients' bowel movements return

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Postacı, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Postaci A, Durgut R, Aytac BG, Ceyhan M. Effect of sugammadex with neostigmine on postoperative bowel function and on recovery of neuromuscular functions: A randomized controlled trial. Medicine (Baltimore). 2024 Sep 13;103(37):e39623. doi: 10.1097/MD.0000000000039623. PMID 39287249